CLINICAL TRIAL: NCT04744844
Title: Does Absence of DNA Amplification in Blastocoel Fluid Enhance Conventional Blastocyst Selection and IVF Outcome?
Brief Title: DNA Amplification in Blastocoel Fluid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for the trial was cancelled by funding organization
Sponsor: Antalya IVF (Other)
Responsible Party: Principal Investigator, Kevin Coetzee, Scientific officer, Antalya IVF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BF 13.1.2021:51
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Clinical Pregnancy; Embryo Implantation
Keywords: DNA; amplification; blastocyst fluid; blastocyst selection; frozen embryo transfer; minimally invasive

STUDY DESIGN:
Intervention Model Description: A single IVF centre double-blind randomised controlled trial.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DNA-amplification selection (Experimental): In the experimental arm, all blastocysts will undergo routine morphological assessment, with the 3 top-scoring blastocysts undergoing blastocoel fluid biopsy (BF-biopsy) and whole-genomic amplification. A single blastocyst with no DNA amplification will be selected for transfer in a frozen embryo transfer cycle.
  Interventions: Procedure: blastocoel fluid biopsy
- Morfological-score selection (Active Comparator): In the active comparator arm, all blastocysts will undergo routine morphological assessment. The (single) top-scoring blastocyst will be selected for transfer in a frozen embryo transfer cycle.
  Interventions: Procedure: blastocoel fluid biopsy

INTERVENTIONS:
Procedure: blastocoel fluid biopsy — In the present study, blastocoel fluid biopsy (BF-biopsy) and collapse will be performed using a microinjection pipette similar to that used to perform ICSI. The pipette will be pushed gently through the zona pellucida and TE, and up to 90% of the BF will be aspirated.

SUMMARY:
Introduction: Although innovative procedural changes in frozen embryo transfer (FET) cycles have increased the implantation rate of blastocysts transferred significantly, blastocyst selection remains a significant limiting factor in implantation outcomes. To improve implantation rates requires conventional microscopic blastocyst morphology scoring/selection technique to be replaced by an enhanced blastocyst selection technique or for the conventional morphology selection technique to be strengthened by novel supplementary selection techniques. Blastocoel fluid biopsy with DNA amplification is a minimally invasive (mi) technique that may supplement a blastocyst morphology score variables with a genetic variable.

Objective: In the present randomized controlled trial (RCT), DNA amplification in blastocoel fluid biopsies (BF-biopsy) will be investigated as a supplementary measure to select blastocysts for transfer in conjunction with blastocyst morphology scores. The objective will be to develop a minimally invasive blastocyst selection technique, which will improve selection and increase clinical implantations, while not increasing costs.

Materials and Methods: A single IVF centre double-blind randomised controlled trial, with patients recruited having female age 18 to 35 years from infertile patients presenting for freeze-all-IVF treatment. Enrolled patients (N = 500) with ≥five 2PN zygotes after ICSI will be randomised (1:1) to the two arms of the trial (i.e., test and control arm). In the test arm, 3 blastocysts will undergo blastocoel fluid biopsy (BF-biopsy) and whole-genomic amplification. Single blastocysts with no DNA amplification will be transferred in FETs of the test arm and single top-scoring blastocysts will be transferred in FETs of the control arm. The primary outcome measure of the trial will be clinical implantation (i.e., gestational sac with fetal heartbeat).

Results: The clinical implantation outcomes of FETs in which score-selected single blastocyst with no DNA amplification and score-selected single blastocysts were transferred will be compared.

DETAILED DESCRIPTION:
Introduction The goal of assisted reproductive technology (ART) is the delivery of a healthy singleton, with the treatment strategy in IVF having the best chance being the transfer of the single most viable embryo from a patient's embryo cohort. Embryo selection, therefore, is paramount to the success of this goal. The microscopic assessment and scoring of embryo morphology was developed as an embryo selection technique in the early years of IVF (Veeck, 1991) and has ever since remained the most widely practised embryo selection technique. However, the technique's limited ability to maximise embryo implantation rates has for long been lamented and, therefore, more enhanced embryo selection techniques have for long been sought. Time-lapse monitoring and scoring (Paulson et al., 2018) and euploid embryo transfer using PGT-A (preimplantation genetic testing for aneuploidy; Gleicher et al., 2017) are recent innovations that have become contenders to replace conventional microscopic assessment and scoring of embryo morphology. An advantage of PGT-A is its independence of embryo development and morphological feature assessments, as euploid blastocysts implant at the same rate irrespective of blastocyst morphology score (Capalbo et al., 2014). Moreover, besides PGT-A's technical and biological limitations, the costs of implementation PGT-A as an embryo selection technique may be regarded prohibitive by many.

In the evolution of PGT in human IVF, PGT has progressed from PGT-v1 to PGT-v2 based on the adverse outcomes of biopsying 1-2 blastomeres from cleavage-stage embryos (PGT-v1) and the improvement in blastocyst development conditions. The evidence suggested that PGT-v.1 posed a significant risk to embryo viability, with no benefit resulting from the transfer of euploid embryos (Gleicher et al., 2017). The majority of studies have reported that PGT-v2, which requires the biopsying of 5-10 trophectoderm (TE) cells, poses no significant risk to the developmental potential (implantation viability) of biopsied blastocysts. However, recently there have been reports, suggesting that TE biopsy may not be completely free of risk (Gleicher et al., 2017, Ozgur et al., 2019). Currently, PGT-A faces four challenges preventing its routine use as a blastocyst selection technique; (1) the need for high technical expertise, (2) the invasiveness of TE biopsy, (3) the cost of the full technique, and (4) that TE biopsy is subject to sampling bias - a single TE biopsy of 5-10 cells may not accurately represent the ploidy of the whole blastocyst.

A spin-off of conventional PGT is the analysis of DNA in blastocoel fluid (BF). This phenomenon was first reported by Palini et al. (2013). The origin of the DNA in BF has been suggested to be the result of embryo euploidisation, i.e., the elimination of aneuploidy DNA or aneuploidic cells through regulatory processes such as apoptosis and or necrosis (Leaver and Wells, 2019). The practice of blastocyst collapse before vitrification (Mukaida et al., 2006, Iwayama et al., 2011) provides the opportunity to perform minimally invasive PGT-A (miPGT-A), i.e., the biopsying BF. In a study to investigate ploidy concordance between PGT-A with TE biopsy and PGT-A with BF biopsy, the authors found that the clinical pregnancy rate was 77% for blastocysts with no DNA amplification were transferred and 37% for blastocysts with DNA amplification (Magli et al., 2018). The mere accumulation of DNA in the BF, therefore, could be used as a supplementary measure to prioritise blastocysts for transfer. Implementing BF-biopsy and whole-genomic amplification (WGA) as a supplementary selection measure limits/reduces three of PGT-A's main challenges; (1) technical expertise, (2) invasiveness, and (3) costs.

In the present randomized controlled trial (RCT), the investigators will investigate DNA amplification in blastocyst fluid biopsies (BF-biopsy) as a supplementary selection technique to select blastocysts for transfer in conjunction with blastocyst morphology scores. The clinical implantation outcomes of FETs in which score-selected single blastocyst with no DNA amplification and score-selected single blastocysts were transferred will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with female age 18≤35 years on the day of consultation (with the clinician projecting female age to be ≤35 on the day of oocyte retrieval).
* Patients who provide informed consent to participate in the trial and for the use of their anonymized data in research.
* Patients with ≤2 previous IVF treatments.
* Patients predicted to have single blastocyst transfers.

Exclusion Criteria:

* Patients with female age >35 years on the day of consultation.
* Female patients with insulin-dependent diabetes or non-insulin-dependent diabetes mellitus and female patients with gastrointestinal, cardiovascular, pulmonary, liver or kidney disease.
* Female patients with any contraindications or allergies to the drugs used in routine freeze-all-IVF.
* Patients undergoing conventional PGT-A (aneuploidy) or PGT-M (monogenic disorders)
* Patients with less than 5 2-PN zygotes on day 1 of embryo development will be excluded from randomization.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
clinical implantation | Transvaginal ultrasound examinations will be performed after 5 weeks of gestation
  Clinical implantation will be defined as a cycle with an ultrasound confirmed normal gestational sac and heartbeat.

SECONDARY OUTCOMES:
pregnancy | Blood serum pregnancy tests will be performed 9 days after blastocyst transfer
  Pregnancy will be defined as a cycle with an arbitrary serum βHCG level of >30 mIU/mL
ongoing pregnancy | Transvaginal ultrasound examinations will be performed after 12 weeks of gestation
  Ongoing pregnancy will be defined as a cycle with an ultrasound confirmed normal gestational sac and heartbeat.

CONTACTS AND LOCATIONS:
Overall Officials: Kemal Ozgur, MD, Study Director — Antalya IVF; Kevin Coetzee, PhD, Principal Investigator — Antalya IVF
Locations (1):
- Antalya IVF, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The IPD plan sharing plan:
  The protocol will be published (word document) on the completion of registration on ClinicalTrials.gov The relevant clinical data will be published on journal acceptance of the study (excel spreadsheet)
Supporting Information: Study Protocol, CSR
Time Frame: To be published immediately after publication acceptance.
Access Criteria: Open access at the Mendeley Data at the URLs provided

REFERENCES:
- [Result] Capalbo A, Rienzi L, Cimadomo D, Maggiulli R, Elliott T, Wright G, Nagy ZP, Ubaldi FM. Correlation between standard blastocyst morphology, euploidy and implantation: an observational study in two centers involving 956 screened blastocysts. Hum Reprod. 2014 Jun;29(6):1173-81. doi: 10.1093/humrep/deu033. Epub 2014 Feb 26. PMID 24578475
- [Result] Iwayama H, Hochi S, Yamashita M. In vitro and in vivo viability of human blastocysts collapsed by laser pulse or osmotic shock prior to vitrification. J Assist Reprod Genet. 2011 Apr;28(4):355-61. doi: 10.1007/s10815-010-9522-4. Epub 2010 Dec 9. PMID 21152966
- [Result] Magli MC, Albanese C, Crippa A, Tabanelli C, Ferraretti AP, Gianaroli L. Deoxyribonucleic acid detection in blastocoelic fluid: a new predictor of embryo ploidy and viable pregnancy. Fertil Steril. 2019 Jan;111(1):77-85. doi: 10.1016/j.fertnstert.2018.09.016. Epub 2018 Dec 5. PMID 30528055
- [Result] Ozgur K, Berkkanoglu M, Bulut H, Yoruk GDA, Candurmaz NN, Coetzee K. Single best euploid versus single best unknown-ploidy blastocyst frozen embryo transfers: a randomized controlled trial. J Assist Reprod Genet. 2019 Apr;36(4):629-636. doi: 10.1007/s10815-018-01399-1. Epub 2019 Jan 7. PMID 30617927
- [Result] Palini S, Galluzzi L, De Stefani S, Bianchi M, Wells D, Magnani M, Bulletti C. Genomic DNA in human blastocoele fluid. Reprod Biomed Online. 2013 Jun;26(6):603-10. doi: 10.1016/j.rbmo.2013.02.012. Epub 2013 Mar 13. PMID 23557766
- [Result] Veeck LL: Atlas of the Human Oocytes and Early Conceptus. 1991, Vol. 2. Baltimore, Williams & Willkins Co.
- [Result] Paulson RJ, Reichman DE, Zaninovic N, Goodman LR, Racowsky C. Time-lapse imaging: clearly useful to both laboratory personnel and patient outcomes versus just because we can doesn't mean we should. Fertil Steril. 2018 Apr;109(4):584-591. doi: 10.1016/j.fertnstert.2018.01.042. No abstract available. PMID 29653705
- [Result] Gleicher N, Metzger J, Croft G, Kushnir VA, Albertini DF, Barad DH. A single trophectoderm biopsy at blastocyst stage is mathematically unable to determine embryo ploidy accurately enough for clinical use. Reprod Biol Endocrinol. 2017 Apr 27;15(1):33. doi: 10.1186/s12958-017-0251-8. PMID 28449669
- [Result] Mukaida T, Oka C, Goto T, Takahashi K. Artificial shrinkage of blastocoeles using either a micro-needle or a laser pulse prior to the cooling steps of vitrification improves survival rate and pregnancy outcome of vitrified human blastocysts. Hum Reprod. 2006 Dec;21(12):3246-52. doi: 10.1093/humrep/del285. Epub 2006 Aug 26. PMID 16936299